CLINICAL TRIAL: NCT07197203
Title: Comparison of Caudal Block and Sacral Erector Spinae Plane Block With Dexmedetomidine in Pediatric Penile Hypospadias Repair
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nancy Makram Gaballah, Residant doctor at Assiut university hospital, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CB VS SESPB Dexmedetomidine
Record Dates: First submitted 2025-09-20; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Hypospadias
MeSH Terms: conditions — Hypospadias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A (Active Comparator): Caudal Epidural Block
  Interventions: Procedure: Caudal epidural block
- Group B (Active Comparator): Sacral ESP Block
  Interventions: Procedure: Sacral ESP Block

INTERVENTIONS:
Procedure: Sacral ESP Block — * Position: Prone with a pillow under the pelvis.
  * Ultrasound: High-frequency linear probe placed parasagittal, 1-1.5 cm lateral to the midline at S2-S3. Structure identified: skin → subcutaneous tissue → erector spinae muscle → sacral lamina.
  * Technique: An echogenic 22G needle will be advanced in-plane until contact with the sacral lamina under the erector spinae muscle. After hydro dissection with saline, the study drug will be injected with visible spread along the fascial plane. The same procedure will be repeated contralaterally.
  * Dose: Bupivacaine 0.25% total 1 mL/kg divided equally on both sides, dexmedetomidine 1 μ g/kg divided equally.
  Arms: Group B
Procedure: Caudal epidural block — * Position: Prone with a pillow under the pelvis.
  * Ultrasound: High-frequency linear probe placed parasagittal, 1-1.5 cm lateral to the midline at S2-S3. Structure identified: skin → subcutaneous tissue → erector spinae muscle → sacral lamina.
  * Technique: An echogenic 22G needle will be advanced in-plane until contact with the sacral lamina under the erector spinae muscle. After hydro dissection with saline, the study drug will be injected with visible spread along the fascial plane. The same procedure will be repeated contralaterally.
  * Dose: Bupivacaine 0.25% total 1 mL/kg divided equally on both sides, dexmedetomidine 1 μ g/kg divided equally.
  Arms: Group A

SUMMARY:
Hypospadias is one of the most common congenital anomalies in childhood, requiring surgical reconstruction (1). It is a penile malformation with a more proximal or ventral location beyond the usual localization of the urethra. Hypospadias is a common congenital urogenital anomaly in male children, and its incidence is reported to be approximately one in every 300 births. However, it is suggested that hypospadias may increase in developed countries (2, 3). Postoperative pain management followinghypospadias repair is of great importance, as inadequatepain control may lead to adverse endocrine, metabolic, and inflammatory stress responses, resulting in higher morbidity and poor recovery(4).

Regional anesthesia has gained increasing attention in pediatric surgery as a valuable tool for managing perioperative pain and improving surgical outcomes(5). The caudal epidural block has long been considered the gold standard technique fo infraumbilical surgeries, including hypospadias repair, due to its proven efficacy and safety (4). However, its limitations include a relatively short durationof analgesia, the need for larger local anesthetic volumes, and potential adverse effects such as motor block, urinary retention, and inadvertent dural puncture. These drawbacks have led anesthesiologists to explore alternative regional techniques(6-8) Recently, the sacral erector spinae plane (ESPB) block has been introduced as a novel technique for postoperative analgesia in children(9, 10). It is an emerging regional anesthetic technique with significant potential for clinical benefit Nevertheless, its exact mechanism(s) of action have been much debated. These mechanisms include neural blockade and central inhibition from direct spread of local anesthetic to the paravertebral or epidural space, and analgesia mediated by elevated local anesthetic plasma concentrations due to systemic absorption(11).

Evidence suggests sacral ESP block can give excellent analgesia in surgical procedures (12-14). Few studies have examined its use to alleviate acute pain after hypospadias surgery (15, 16). There is a lack of data on the postoperative analgesic efficacy in hypospadias surgery.

The addition of adjuvant agents to local anesthetics has been shown to enhance the quality and duration of regiona anesthesia(17).

Dexmedetomidine, an alpha-2 adrenergic agonist, has gained significant attention for its sedative, analgesic, and anxiolytic properties in pediatric anesthesia(18).

Dexmedetomidine, a highly selective α 2- α 2-adrenergic agonist, has demonstrated sedative and analgesic properties without significant respiratory depression, making it particularly attractive in pediatric anesthesia. When used as an adjuvan to local anesthetics, dexmedetomidine prolongs block duration and reduces rescue analgesic requirements(17).

Despite the established role of caudal block and the emerging potential of sacral ESPB, there is a lack of randomized controlled trials directly comparing their analgesic efficacy in pediatric patients when combined with dexmedetomidine

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients, aged 1-6 years, ASA physical statusI- II, scheduled for elective hypospadias repair surgery under general anesthesia.

Exclusion Criteria:

* • Parental refusal.

  * Allergy to local anesthetics or dexmedetomidine.
  * Coagulation disorders.
  * Local infection at the site of injection.
  * Anatomical abnormalities (e.g., spina bifida, sacralmalformations).
  * Neurological disease.

Ages: 1 Year to 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — male
Enrollment: 66 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
postoperative analgesia period | 24 hours
  duration of postoperative analgesia in studied patients